CLINICAL TRIAL: NCT04444453
Title: Early Ambulation to Reduce Hospital Length of Stay
Acronym: EARLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202001410; IRB202001410 (Other: IRB-01)
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Ambulation; Wearable Devices
Keywords: length of stay; hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pedometer (Experimental): Admitted patients who receive a pedometer to wear during their hospital stay to measure steps ambulated
  Interventions: Device: Wearable Pedometer
- Control (No Intervention): Patients admitted to hospital who do not receive a pedometer, but receive all other usual standard of care

INTERVENTIONS:
Device: Wearable Pedometer — Pedometer worn on wrist
  Other Names: Pedometer
  Arms: Pedometer

SUMMARY:
Early ambulation of inpatients has been shown to be a key driver of decreased LOS and also reduced adverse events such as venous thromboembolism (VTE). We will test if a patient wearable device (pedometer) measuring steps and ambulation sessions decreases hospital LOS (primary outcome), decreases hospital LOS index (LOSI), decreases time to first ambulation, decreases time to first bowel movement (BM), decreases incidence of VTEs, and decreases costs (secondary outcomes). In a pilot randomized control trial, we will randomize 150 total adult patients admitted to UF Health Jacksonville in a 1:1 fashion to usual care and wearable pedometer or usual care. Patients randomized to the study intervention will receive a wearable pedometer upon admission, to be worn for the duration of their inpatient stay. Study outcome measures to be compared between the pedometer and no pedometer group include hospital LOS (primary outcome), hospital LOSI, time to first ambulation, time to first BM, incidence of VTEs, patient experience, and costs (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages > or equal to 18 years
2. Patient has capacity to undergo informed consent
3. Admitted to UF Health Jacksonville 8N progressive inpatient unit
4. Inpatient physician orders for patient ambulation and/or activity as tolerated upon hospital admission
5. Patient with a Fall Predictive Analytics score category of "low risk"
6. Patient with a Morse Fall Scale (MFS) of < or equal to 50
7. No contraindications to wearing a wrist pedometer (no skin breakdown, overlying skin infections, contact dermatitis, or indwelling catheters/need for venipuncture at wrist site)

Exclusion Criteria:

1. Patient < 18 years of age
2. Patient without capacity to undergo informed consent
3. Patient with a 'do not ambulate' order or has order for bed rest or other contraindication to ambulation (i.e., fall risk) or dependent on more than minimal assistance to ambulate
4. Patient with a Fall Predictive Analytics score category of "high risk"
5. Patient with MFS > 50 or labelled by clinical team as fall risk
6. Non-English speaking
7. In law enforcement custody or ward of the state
8. Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | Up to 1 month
  Time patient is admitted in hospital

SECONDARY OUTCOMES:
Hospital length-of-stay index | Up to 1 month
Time to first ambulation | Up to 1 month
Time to first bowel movement | Up to 1 month
Rate of venous thromboembolism | Up to 1 month
Total hospitalization costs | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fishe, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No